CLINICAL TRIAL: NCT04071067
Title: Anemia of Inflammation and Deficiency Anemia in Critically Ill Patients; Biological Markers
Brief Title: Anemia of Inflammation and Deficiency Anemia
Acronym: AIDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Constantin Bodolea, Head of 2nd Anesthesia Department, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 89/8.04.2019
Record Dates: First submitted 2019-07-01; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Anemia, Iron Deficiency; Anemia of Chronic Disease
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency Clinical County Hospital Group
- Municipal Clinical Hospital Group

SUMMARY:
Critical patients which requiring admission to intensive care (IT) are a special group of patients. In these patients the prevalence of anemia reported in studies is 75%. This prevalence is similar to that in the retrospective observational study conducted in our intensive care unit(ICU). Of the 783 patients included in the study, 551 (73.37%) had anemia on admission. Frequently anemia is present on discharge from ICU or hospital and may persist for an average of 11 weeks. Some studies have reported the presence of anemia as far as 6 months after discharge. It is widely accepted that anemia has a negative impact on rehabilitation and quality of life, but the treatment can not be exclusively based on blood products due to the risks associated with transfusion. Alternative treatments such as injectable iron or erythropoietin should be considered.

The Transfusion Management Initiative Group recently issued recommendations on perioperative anemia. Similar recommendations for ICU have not yet been developed in Romania. The current study has two main purposes. The first to adopt the perioperative anemia diagnostic algorithm and adapt it to anemic patients on ICU; the second to identify patients with mixed anemia (inflammatory and iron deficient anemia) who can benefit from treatment with iron.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to ICU

ICU stay >48hours

Exclusion Criteria:

* Refusal to participate in the study
* Allergy to iron products
* Anemia requiring massive transfusion in the last 7 days
* Treatment of iron products in the last 7 days
* Chronic renal failure with GFR <30mL / min or on dialysis
* Metabolism of iron
* Pregnant or lactation patients
* Rheumatic diseases
* Inflammatory bowel diseases
* Hematological pathologies
* Impossibility of performing laboratory tests within 72 hours of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU during the study period which do not meet any exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin levels during ICU stay | 21 days: day 0=point 1; day 7=point 2; day 14=point 3; day 21 =point 4;
Number of transfusions during ICU stay | Up to 3 months of hospital stay

SECONDARY OUTCOMES:
Days spent on ICU | Up to 3 months of hospital stay
Days spent in hospital | Up to 3 months
Change in hemoglobin level during hospital stay | Up to 3 months: week 3=point 1; week 6=point 2; week 9=point 3; week 12=point4
Number of hours of mechanical ventilation during hospital stay | Up to 3 months

OTHER OUTCOMES:
Change in hepcidin levels | Days 0, 3, 7, 14, 21
  Hepcidin is a peptide produced by the liver. It acts by binding to ferroportin, the sole exporter of iron. The hepcidin-ferroportin complex is sequestrated in the cytosol of cells followed by its degradation. Ferroportin degradation prevents iron from being exported from the cell.

CONTACTS AND LOCATIONS:
Overall Officials: Constantin Bodolea, Md PhD, Principal Investigator — 2nd Anesthesia Department of University of Medicine and Pharmacy Cluj Napoca
Locations (2):
- Romania (2):
  - Emergency Clinical County Hospital Cluj Napoca, Cluj-Napoca, Cluj
  - Municipal Clinical Hospital Cluj, Cluj-Napoca, Cluj

REFERENCES:
- [Background] Filipescu D, Banateanu R, Beuran M, Burcos T, Corneci D, Cristian D, Diculescu M, Dobrota A, Droc G, Isacoff D, Gosa D, Grintescu I, Lupu A, Mirea L, Posea C, Stanca O, Stefan M, Tomescu D, Tudor C, Ungureanu D, Mircescu G. Perioperative Patient Blood Management Programme. Multidisciplinary recommendations from the Patient Blood Management Initiative Group. Rom J Anaesth Intensive Care. 2017 Oct;24(2):139-157. doi: 10.21454/rjaic.7518.242.fil. PMID 29090267